CLINICAL TRIAL: NCT06710977
Title: A Double-blind, Randomized Controlled Pilot Study Comparing the Safety and Efficacy of Intracameral Levofloxacin and Intracameral Cefazolin in Cataract Surgery
Brief Title: To Compare the Safety and Efficacy of Intracameral Levofloxacin and Intracameral Cefazolin in Reducing Rates of Endophthalmitis Following Cataract Surgery.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021/00844-SSR3
Record Dates: First submitted 2024-11-20; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safety of Intracameral levofloxacin in cataract surgery (Experimental): Eligible and recruited patients are randomized to intracameral levofloxacin or intracameral cefazolin during cataract surgery
  Interventions: Drug: Safety of intracameral levofloxacin in cataract surgery; Drug: Use of intracameral cefazolin in cataract surgery
- Use of intracameral cefazolin in cataract surgery (Active Comparator): Eligible and recruited patients were randomized to intracameral levofloxacin or intracameral cefazolin during cataract surgery
  Interventions: Drug: Safety of intracameral levofloxacin in cataract surgery; Drug: Use of intracameral cefazolin in cataract surgery

INTERVENTIONS:
Drug: Safety of intracameral levofloxacin in cataract surgery — Intracameral levofloxacin (0.1ml/0.5mg)
Drug: Use of intracameral cefazolin in cataract surgery — Intracameral cefazolin (0.1ml/1mg)

SUMMARY:
Patients with senile cataracts undergoing phacoemulsification were assigned to receive intracameral levofloxacin (0.1ml/0.5mg) or intracameral cefazolin (0.1ml/1mg). The primary endpoint was the occurrence of endophthalmitis during the 3 month follow-up period. Secondary endpoints included best-corrected visual acuity (BVCA), the presence of anterior chamber (AC) inflammation with grading of AC cells and presence of flare, along with intraocular pressure (IOP), corneal cell thickness (CCT), central foveal thickness (CFT) and cell density.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥50 to <80 years
* Undergoing cataract surgery under the care of one of three study investigators, all of whom were consultant level cataract surgeons
* Only those with senile cataracts, assessed using the Lens Opacities Classification System III scale (LOCS III) and without features of complex cataracts were included

Exclusion Criteria:

* <50 or >80 years old
* Prior ocular trauma, pregnant, previous history of refractive, corneal or intraocular surgery, cornea endothelial cell count <1500/sqmm², concomitant ocular disease, allergy to penicillin, fluoroquinolone or cephalosporin, and abnormal biometric measurements

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment related adverse events to Intracameral Cefazolin versus Levofloxacin | From cataract surgery through to study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - Ang Mo Kio Specialist Center, Singapore

IPD SHARING:
Plan to Share IPD: No
Upon publication, we will be providing contact details such that keen parties can approach us to get clarification or access to the data.

REFERENCES:
- [Background] Cruz FM, Uy HS, Rubio CJ, Chan PS. Postoperative Safety Outcomes in Patients Undergoing Routine Phacoemulsification Cataract Surgery with Intraoperative Intracameral Injection of Preservative-Free Moxifloxacin versus Levofloxacin. Philippine Journal of Ophthalmology. 2022;47(1)
- [Background] Espiritu CRG, Bolinao JG. Prophylactic intracameral levofloxacin in cataract surgery - an evaluation of safety. Clin Ophthalmol. 2017 Dec 12;11:2199-2204. doi: 10.2147/OPTH.S144625. eCollection 2017. PMID 29276375
- [Derived] Koh YT, Yeo TK, Toh ZH, Wong JXH, Ngo WK, Fam HB, Pek DCK. A double-blind, randomized controlled pilot study comparing the safety of intracameral levofloxacin and intracameral cefazolin in patients undergoing cataract surgery. Sci Rep. 2025 Oct 2;15(1):34444. doi: 10.1038/s41598-025-17553-6. PMID 41038947